CLINICAL TRIAL: NCT06541821
Title: Investigation of Physical Activity, Kinesiophobia, and Stoma Compliance in Patients Undergoing Urostomy for Bladder Cancer
Brief Title: Physical Activity, Kinesiophobia, and Stoma Compliance in Urostomy Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Assist. Prof. Dr., Selcuk University
Other Study IDs: 2024/07.25
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urostomy Patients Group
  Interventions: Other: survey evaluation
- Control Group
  Interventions: Other: survey evaluation

INTERVENTIONS:
Other: survey evaluation — assessment of physical activity, fear of movement, and ostomy compliance

SUMMARY:
In this study, it is aimed to determine the level of physical activity, to investigate kinesiophobia, to determine compliance with the stoma and to compare with healthy controls in patients with bladder cancer who have undergone urostomy surgery and live with a stoma.

ELIGIBILITY:
Inclusion Criteria:

* The patient group will include people between the ages of 40-75 who underwent urostomy surgery and a stoma after being diagnosed with bladder cancer.
* The control group will include age-matched healthy people with similar age, body weight and height, without a previous history of cancer.

Exclusion Criteria:

* Orthotopic surgeries will not be included in the patient group
* Being under the age of 40,
* Being diagnosed with lymphedema,
* Presence of active metastasis,
* Neurological pathologies that limit voluntary mobility,
* Orthopedic and cardiovascular pathologies,
* Having a learning disability or other cognitive or communication impairment.
* The control group will be excluded if they have any history of cancer.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients using ostomy after Urostomy Surgeries for Bladder Cancer
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-02 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire Short Form (IPAQ-SF) | 10 minutes
  To assess physical activity levels in METs
Tampa Kinesiophobia Scale | 10 minutes
  assess fear of movement in patients
Ostomy Compliance Scale | 10 minutes
  Determination of psychosocial adaptation levels of individuals with ostomy to ostomy

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selçuklu, Turkey (Türkiye)